CLINICAL TRIAL: NCT03245307
Title: A Single-center, Open-Label, Drug Interaction Study to Determine the Effects of Apatinib on the Metabolism of CYP3A4/5 and CYP2C9 Probe Drugs in Patients With Solid Tumors
Brief Title: A Study To Test The Effect Of Apatinib On P450 Enzymes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-APTN-DDI-01
Record Dates: First submitted 2017-07-17; First posted 2017-08-10 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2017-07

CONDITIONS: Cytochrome P450 Interaction
MeSH Terms: interventions — apatinib; Nifedipine; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treament (Experimental): In phase A, subjects receiving a single 30 mg oral dose of Nifedipine controlled-release tablets and wash-out for 2 days,a single 3 mg oral dose of warfarin tablets and wash-out for 12 days, then apatinib 750 mg once daily with a single 30 mg oral dose of Nifedipine controlled-release tablets co-administered on day 6 ,a a single 3 mg oral dose of warfarin tablets co-administered on day 9.
  Interventions: Drug: Apatinib; Drug: Nifedipine GTIS; Drug: Warfarin Potassium

INTERVENTIONS:
Drug: Apatinib — Apatinib at a dosage of 750mg will be administered daily from day 9 of phase A
Drug: Nifedipine GTIS — Nifedipine at a dosage of 30mg will be administered at day 1 and day 14 of phase A
  Other Names: Nifedipine
Drug: Warfarin Potassium — Nifedipine at a dosage of 3mg will be administered at day 3 and day 16 of phase A
  Other Names: warfarin

SUMMARY:
Apatinib, an oral inhibitor of vascular endothelial growth factor receptor 2（VEGFR-2）, inhibits multiple cytochrome P450 (CYP450) enzymes in vitro. This study in patients with advanced cancer evaluated the effect of Apatinib on CYP450 function by comparing the pharmacokinetics of CYP-specific probe drugs in the presence and absence of Apatinib. The probes used included Nifedipine (CYP3A specific), warfarin (CYP2C9 specific).

DETAILED DESCRIPTION:
This open-label study consists of a drug interaction phase that (part A) and a drug-continuation phase (part B). Patients will receive CYP450-probe drugs, and PK assessments will be performed before apatinib-administration and aſter once-daily administration of apatinib for 5 days (the predicted time point when steady-state plasma apatinib concentrations will have been achieved).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumors.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow, renal, lung, and liver function.
* A female subject must not be pregnant and will agree not to become pregnant during the trial

Exclusion Criteria:

* Primary carcinoma of liver
* Any major surgery, chemotherapy, hormone therapy, investigational drugs, or radiotherapy within the last 28 days.
* Poorly controlled hypertension.
* A prior history of cardiovascular disease, arrhythmias, or significant ECG abnormalities, and corrected QT (QTc) prolongation defined as a QTc interval greater than or equal to 450 msec(male) or 470 msec(female).
* Arterial or venous thrombi (including cerebrovascular accident).
* Current use of therapeutic anticoagulation (low molecular weight heparin, oral anticoagulant agents).
* Active brain metastases.
* A history of bleeding problems.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of warfarin or nifedipine | 1 year
  AUC0~t of warfarin and nifedipine in the absence or in presence of apatinib will be defined

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Day 1 to 21 ( Phase A）
  to assess safety and tolerability of apatinib combined with warfarin or nifedipine in patients with advanced solid tumors. The vital signs, ECG, laboratory values and adverse events (AE and SAE) were judged according to NCI-CTCAE V4.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Medical University First Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided